CLINICAL TRIAL: NCT07264660
Title: Diagnostic Value of Transcervical True-Cut Biopsy in Uterine Masses
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma AL_Zahraa Mohamed Mokhtar, Dr, Assiut University
Other Study IDs: Biopsy in Uterine Masses
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Uterine Tumor
MeSH Terms: conditions — Uterine Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1
  Interventions: Procedure: Transcervical True-Cut Biopsy

INTERVENTIONS:
Procedure: Transcervical True-Cut Biopsy — Transcervical True-Cut Biopsy in Uterine Masses

SUMMARY:
Uterine tumor-like masses represent a wide spectrum of gynecological conditions, ranging from benign lesions such as myomas and adenomyosis to malignant tumors like endometrial carcinoma and leiomyosarcoma, as well as other entities including gestational trophoblastic disease [4]. Accurate preoperative diagnosis is crucial, since management varies from conservative follow-up to radical surgery or systemic therapy.

Imaging modalities such as ultrasound and MRI are essential in the initial evaluation of uterine masses, providing information on size, location, and internal characteristics. However, imaging alone often lacks specificity, as benign and malignant lesions may share overlapping features [4]. Thus, histopathological confirmation remains the gold standard.

Among available diagnostic approaches, transcervical ultrasound-guided true-cut biopsy offers unique advantages. Unlike dilatation and curettage, which may yield insufficient or fragmented tissue, this technique retrieves core samples with preserved architecture [1]. Compared to hysteroscopic biopsy, which mainly targets endometrial lesions and frequently requires anesthesia, the transcervical route can access intramural and submucosal lesions in a simple outpatient setting [2]. While Novak biopsy is suitable for outpatient endometrial sampling, it cannot adequately reach deeper myometrial or submucosal masses [4]. Furthermore, unlike the transabdominal approach, which may be limited by bowel interposition or patient habitus, the transcervical technique ensures direct, real-time ultrasound-guided targeting with high feasibility and accuracy [3].

Preliminary studies have demonstrated high sensitivity and specificity for transcervical true-cut biopsy [1-3,5]. However, prior research was often limited by small sample sizes, focus on specific pathologies rather than the full spectrum of uterine tumor-like masses, and lack of direct comparison with excisional biopsy as a gold standard. Therefore, this study will assess its diagnostic value in scheduled patients with uterine tumor-like masses, by evaluating the agreement between transcervical biopsy results and excisional biopsy. Ultimately, the aim is to determine whether this minimally invasive, outpatient technique can help avoid unnecessary surgeries in benign cases and ensure that patients with malignant disease proceed promptly to the most appropriate surgical intervention

ELIGIBILITY:
Inclusion Criteria:

* • Women diagnosed with uterine tumor-like masses by imaging and scheduled for surgical excision.

  * Non-virgin patients .

Exclusion Criteria:

* • Patients with active genital tract infection.

  * Patients with bleeding disorders or on uncorrected anticoagulation therapy.
  * .Pregnancy.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: • Women diagnosed with uterine tumor-like masses by imaging and scheduled for surgical excision
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
• Diagnostic accuracy of transcervical ultrasound-guided true-cut biopsy compared to the gold standard excisional biopsy | 1 year
  • Diagnostic accuracy of transcervical ultrasound-guided true-cut biopsy compared to the gold standard excisional biopsy

REFERENCES:
- [Background] Park JJ, Kim CK, Park BK. Ultrasound-Guided Transvaginal Core Biopsy of Pelvic Masses: Feasibility, Safety, and Short-Term Follow-Up. AJR Am J Roentgenol. 2016 Apr;206(4):877-82. doi: 10.2214/AJR.15.15702. Epub 2016 Feb 25. PMID 26913556
- [Background] Asp M, Mockute I, Masback A, Liuba K, Kannisto P, Malander S. Tru-Cut Biopsy in Gynecological Cancer: Adequacy, Accuracy, Safety and Clinical Applicability. J Multidiscip Healthc. 2023 May 15;16:1367-1377. doi: 10.2147/JMDH.S396788. eCollection 2023. PMID 37215751
- [Background] Quintana-Berto R, Padilla-Iserte P, Gil-Moreno A, Oliver-Perez R, Coronado PJ, Martin-Salamanca MB, Pantoja-Garrido M, Lorenzo C, Beric D, Gilabert-Estelles J, Sanchez L, Roldan-Rivas F, Diaz-Feijoo B, Rodriguez-Hernandez JR, Marcos-Sanmartin J, Muruzabal JC, Canada A, Domingo S; SEGO Spain-GOG Group. Preoperative sampling in endometrial cancer: evaluation of the histopathological agreement with definitive surgical specimen. Clin Transl Oncol. 2022 Dec;24(12):2388-2394. doi: 10.1007/s12094-022-02893-w. Epub 2022 Aug 19. PMID 35984612
- [Background] Asaturova A, Zaretsky A, Rogozhina A, Tregubova A, Badlaeva A. Advancements in Minimally Invasive Techniques and Biomarkers for the Early Detection of Endometrial Cancer: A Comprehensive Review of Novel Diagnostic Approaches and Clinical Implications. J Clin Med. 2024 Dec 11;13(24):7538. doi: 10.3390/jcm13247538. PMID 39768459